CLINICAL TRIAL: NCT02376361
Title: Hemodialysis Access Surveillance Evaluation Study
Acronym: HASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Transonic Systems Inc. (Industry)
Responsible Party: Principal Investigator, Loay Salman, MD, Professor of Medicine, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20140235
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Hemodialysis Access; Thrombosis
Keywords: Surveillance
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surveillance Group (Active Comparator): Monthly blood flow surveillance by ultrasound dilution technique and standard of care.
  Interventions: Device: Transonic
- Control Group (No Intervention): Control group will receive standard monitoring (standard care).

INTERVENTIONS:
Device: Transonic — Access recirculation, access flow would be determined using the ultrasound dilution technique (Transonic system).
  1. Within 90 min of the beginning of HD session HD03 sensors are clamped HD tubing lines
  2. Recirculation, access flow will be performed according to HD03 Manual.
  3. Post intervention evaluation is as per each arm follow up unless other follow up deemed necessary by the interventionalist.
  Arms: Surveillance Group

SUMMARY:
The purpose of the study is to learn if monitoring dialysis access blood flow during dialysis treatment with a transonic machine (an ultrasound technique) will prevent (or reduce) the development of dialysis access thrombosis (clotting).

Investigators would like to study if monitoring with a specific technique called ultrasound dilution technique can help prevent problems with access when compared to what is the current standard of care for patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients undergoing dialysis therapy via an upper extremity arteriovenous access (arteriovenous fistula or an arteriovenous graft) will be enrolled to have monthly surveillance flow measurement using Transonic system or physical examination of the arteriovenous access by qualified person at least once a month for a period of 2 years.

Exclusion Criteria:

* Patients requiring surgical intervention on the arteriovenous access.
* History of access thrombosis (one or more access thrombosis of the current arteriovenous access).
* Patients with signs of access infection.
* Patients with a malignancy.
* Patients with life expectancy of less than six months.
* Unable to understand the study.
* Unable to sign the consent form.
* Patients with psychiatric disorder.
* Age less than 18 or greater than 80 years.
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loay Salman, MD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - North America Research Institute, Azusa, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Albany Medical College, Albany, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Surveillance Group: Monthly blood flow surveillance by ultrasound dilution technique and standard of care.
  Transonic: Access recirculation, access flow would be determined using the ultrasound dilution technique (Transonic system).
  1. Within 90 min of the beginning of HD session HD03 sensors are clamped HD tubing lines
  2. Recirculation, access flow will be performed according to HD03 Manual.
  3. Post intervention evaluation is as per each arm follow up unless other follow up deemed necessary by the interventionalist.
Period: Overall Study
Arm/Group | Surveillance Group | Control Group
Started | 229 | 207
Completed | 58 | 90
Not Completed | 171 | 117

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surveillance Group | Control Group | Total
Number analyzed (Participants) | 229 | 207 | 436
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 132 | 108 | 240
  >=65 years | 97 | 99 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.996 (11.855) | 61.826 (11.942) | 61.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 76 | 156
  Male | 149 | 131 | 280
Race/Ethnicity, Customized [Number; unit: participants]
  black | 43 | 43 | 86
  Hispanic | 136 | 93 | 229
  White | 40 | 61 | 101
  Asian/Pacific Islander | 8 | 5 | 13
  Not reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 229 | 207 | 436

OUTCOME MEASURES:

1. Primary Outcome: Hemodialysis Access Thrombosis Rate
Description: Evaluate the reduction of hemodialysis access thrombosis rate
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: thrombotic events per patient
Arm/Group | Surveillance Group | Control Group
Number analyzed (Participants) | 229 | 207
thrombotic events per patient | 0.122 [0.081 to 0.177] | 0.227 [0.167 to 0.302]

2. Secondary Outcome: Tunneled Hemodialysis Catheter Rate
Description: Evaluate the reduction of tunneled hemodialysis catheter rate
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: Events per patient
Arm/Group | Surveillance Group | Control Group
Number analyzed (Participants) | 229 | 207
Events per patient | 0.039 [0.018 to 0.075] | 0.053 [0.027 to 0.095]

3. Secondary Outcome: Number of Participants With a Tunneled Hemodialysis Catheter
Time Frame: Up to 24 months
Measure: Number; unit: participants
Arm/Group | Surveillance Group | Control Group
Number analyzed (Participants) | 229 | 207
participants | 9 | 11

4. Secondary Outcome: Number of Hemodialysis Access Thrombectomy Procedures
Description: Evaluate the reduction of hemodialysis access thrombectomy procedures
Time Frame: Up to 24 months
Measure: Number; unit: Procedures
Arm/Group | Surveillance Group | Control Group
Number analyzed (Participants) | 229 | 207
Procedures | 28 | 47

5. Secondary Outcome: Number of Hemodialysis Access Angiogram and Angioplasty Procedures
Description: Evaluate the reduction of hemodialysis access angiogram and angioplasty procedures
Time Frame: Up to 24 months
Measure: Number; unit: Procedures
Arm/Group | Surveillance Group | Control Group
Number analyzed (Participants) | 229 | 207
Procedures | 227 | 203

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Surveillance Group: Monthly standard of care and blood flow surveillance for the duration of the study
- Control Group: Monthly standard of care for the duration of the study
Arm/Group | Surveillance Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/229 | 0/207
Serious Adverse Events (participants affected / at risk) | 0/229 | 0/207
Other Adverse Events (participants affected / at risk) | 0/229 | 0/207

LIMITATIONS AND CAVEATS:
Study did not achieve targeted numbers for enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT02376361/Prot_SAP_000.pdf